CLINICAL TRIAL: NCT01007175
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study Of The Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, And Clinical Efficacy Of ATN-103 Administered To Japanese Subjects With Active Rheumatoid Arthritis On A Background Of Methotrexate
Brief Title: Study Evaluating Multiple Ascending Doses Of ATN-103 In Japanese Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3242K1-2001; B2271004
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-01

CONDITIONS: Rheumatoid Arthritis
Keywords: TNF inhibitor; Multiple ascending dose study
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental)
  Interventions: Biological: ATN-103 10 mg q4wks
- Cohort 2 (Experimental)
  Interventions: Biological: ATN-103 30 mg q4wks
- Cohort 3 (Experimental)
  Interventions: Biological: ATN-103 80 mg q4wks
- Cohort 4 (Experimental)
  Interventions: Biological: ATN-103 10 mg q8wks
- Cohort 5 (Experimental)
  Interventions: Biological: ATN-103 80 mg q8wks

INTERVENTIONS:
Biological: ATN-103 10 mg q4wks — ATN-103 160-mg vials (lyophilized) and placebo vials (lyophilized) Each subject will be given a single SC injection (0.1 mL) of either ATN-103 or placebo at 4-week intervals for a total of 4 SC injections.
  Arms: Cohort 1
Biological: ATN-103 30 mg q4wks — ATN-103 160-mg vials (lyophilized) and placebo vials (lyophilized) Each subject will be given a single SC injection (0.3 mL) of either ATN-103 or placebo at 4-week intervals for a total of 4 SC injections.
  Arms: Cohort 2
Biological: ATN-103 80 mg q4wks — ATN-103 160-mg vials (lyophilized) and placebo vials (lyophilized) Each subject will be given a single SC injection (0.8 mL) of either ATN-103 or placebo at 4-week intervals for a total of 4 SC injections.
  Arms: Cohort 3
Biological: ATN-103 10 mg q8wks — ATN-103 160-mg vials (lyophilized) and placebo vials (lyophilized) Each subject will be given a single SC injection (0.1 mL) of either ATN-103 or placebo at 8-week intervals for a total of 2 SC injections.
  Arms: Cohort 4
Biological: ATN-103 80 mg q8wks — ATN-103 160-mg vials (lyophilized) and placebo vials (lyophilized) Each subject will be given a single SC injection (0.8 mL) of either ATN-103 or placebo at 8-week intervals for a total of 2 SC injections.
  Arms: Cohort 5

SUMMARY:
This primary purpose of this study is to evaluate the safety, tolerability, and pharmacokinetic properties of multiple ascending doses of ATN-103 administered subcutaneously (below the skin) to Japanese subjects with active rheumatoid arthritis and on a stable background of methotrexate. Some subjects will receive ATN-103 while other subjects will receive a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Meets the ACR 1987 revised criteria for classification of Rheumatoid Arthritis (RA).
* ACR functional class I through III.
* Active RA at the time of screening and at baseline consisting of = 6 swollen and = 6 tender joints at least.
* hs-CRP level = 8 mg/L.
* Must be receiving MTX for at least 12 wks, with a stable dose and route of MTX for at least 6 wks prior to the baseline and continuing on that dose for the duration of the study.
* The report of a chest x-ray performed within 12 wks before the screening documenting the absence of any evidence of malignancy, infection, or abnormalities suggestive of TB must be obtained and available in the subject's study file prior to baseline.
* All WOCBP must have a negative pregnancy test result at screening and baseline.
* All WOCBP who have sexual intercourse with a nonsurgically sterilized male partner must agree and commit to the use of the following highly effective forms of contraception for the duration of the study and for 8 wks after the last dose of investigational product.
* All male subjects who are biologically capable of fathering children must agree and commit to the use of a reliable method of birth control for the duration of the study and for 8 wks after the last dose of investigational product.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Presence of active infections or open cutaneous ulcers or any underlying disease that could predispose subjects to infections or history of serious infection within 4 wks before the baseline.
* A history or current evidence of latent or active TB, evidence of prior or currently active TB by chest X-ray, recent close contact with an individual with active TB, or a positive Mantoux tuberculin skin test.
* Other significant concurrent medical conditions at the time of the screening or baseline.
* Laboratory abnormalities at screening. Positive for HBsAg, HBcAb, and/or HepCAb. ALTand/or AST= 2 times the ULN or higher. Hemoglobin = 8.5 g/dL or lower. Platelet = 125,000 /mm³ or lower, or = 1,000,000 /mm³ or higher. WBC = 3500 /mm³ or lower. Serum creatinine= 2 mg/dL or higher.
* Any prior use of B cell-depleting therapy.
* Receipt within 24 wks before the baseline visit:

Any cytotoxic drugs. Leflunomide. Any investigational biological drug(s).

* Receipt within 12 wks before the baseline visit: Any biological drugs not listed under the exclusion criteria. Any surgical joint interventions (open or arthroscopic). Any investigational drugs (other than investigational biological drugs), procedures, or devices.
* Receipt within 8 wks before the baseline: Abatacept. Any type of TNF inhibitors not listed under the exclusion criteria.
* Receipt within 4 wks before the baseline: Any DMARDs, other than stable background MTX, or immunosuppressive drugs not listed under the exclusion criteria.
* Etanercept. IA hyaluronic acid injections. Any live (attenuated) vaccine.
* Receipt within 2 wks before the baseline: > 10 mg/day of oral prednisone or equivalent, or change in the dose of oral prednisone or its equivalent.
* IA, bolus IM, or IV treatment with corticosteroids. > 1 NSAID, change of dose of the NSAID, or NSAID use greater than the maximum recommended dose.
* Initiation of statins or dosage adjustment to a current statin. Change in the dose of folic acid.
* Known or suspected allergy to ATN-103, any type of TNF inhibitors, human immunoglobulin proteins, or other compounds related to these classes of medication.
* Current or history of psychiatric disease or alcohol or drug abuse that, in the opinion of the investigator, would interfere with the ability to comply with the study protocol or give informed consent.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be evaluated on the basis of AEs, SAEs,(including injection site reactions and infections), physical examination findings, vital sign, measurements, immunogenicity assessments, early termination, and clinical laboratory test. | 20 weeks

SECONDARY OUTCOMES:
Clinical efficacy for Rheumatoid Arthritis (RA) based on ACR responses, ACR-N, DAS 28 and EULAR response. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Josefin-Beate Holz, Study Director — Ablynx, a Sanofi company
Locations (15):
- Japan (15):
  - Investigational Site, Chiba
  - Investigational Site, Ehime
  - Investigational Site, Fukuoka
  - Investigational Site, Gunma
  - Investigational Site, Hyōgo
  - Investigational Site, Kumamoto
  - Investigational Site, Kyoto
  - Investigational Site, Miyazaki
  - Investigational Site, Nagano
  - Investigational Site, Nagasaki
  - Investigational Site, Osaka
  - Investigational Site, Saga
  - Investigational Site, Saitama
  - Investigational Site, Tokyo
  - Investigational Site, Toyama